CLINICAL TRIAL: NCT03471078
Title: Randomized, Double-Blind, Placebo-Controlled Study With Open-Label Extension to Evaluate the Efficacy and Safety of Avatrombopag for the Treatment of Chemotherapy-Induced Thrombocytopenia in Subjects With Active Non-Hematological Cancers
Brief Title: Avatrombopag for the Treatment of Chemotherapy-Induced Thrombocytopenia in Adults With Active Non-Hematological Cancers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sobi, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AVA-CIT-330
Record Dates: First submitted 2018-03-07; First posted 2018-03-20 (Actual); Results first posted 2021-11-24 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chemotherapy-induced Thrombocytopenia
Keywords: CIT; Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia | interventions — avatrombopag

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Avatrombopag (Experimental): Study is 2:1 randomization ratio (avatrombopag to placebo). Investigational product administered orally once daily for 5 days prior to chemotherapy and 5 days following chemotherapy treatment.
  Interventions: Drug: Avatrombopag
- Placebo (Placebo Comparator): Study is 2:1 randomization ratio (avatrombopag to placebo). Investigational product administered orally once daily for 5 days prior to chemotherapy and 5 days following chemotherapy treatment.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Avatrombopag — Oral avatrombopag tablet
  Arms: Avatrombopag
Drug: Placebo Oral Tablet — Placebo comparator tablet
  Arms: Placebo

SUMMARY:
Phase 3 randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of avatrombopag in subjects with chemotherapy-induced thrombocytopenia receiving chemotherapy for the treatment of ovarian, lung (small cell and non-small cell) and bladder cancer.

DETAILED DESCRIPTION:
Subjects will receive placebo controlled test treatment for one cycle of chemotherapy followed by an observational cycle. Subjects will have the option to continue into an open label extension period for all remaining chemotherapy cycles within the current regimen. After the follow-up visit, all subjects will continue to a long-term safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women greater than or equal to 18 years of age;
* A diagnosis of ovarian, lung (small cell or non-small cell) or bladder cancer requiring systemic chemotherapy
* Participant receiving a chemotherapy regimen given in a 21 or 28-day cycle, including 1 or more of the following agents or class of agents:

  * Nucleoside analog, including gemcitabine and fluorouracil;
  * Carboplatin or cisplatin;
  * Anthracycline; or
  * Alkylating agent;
* Participant experienced severe thrombocytopenia, defined as 2 platelet counts <50 x 109/L measured at least 24 hours apart, during the qualifying chemotherapy cycle, of their current chemotherapy regimen
* ECOG performance status <=2

Exclusion Criteria:

* Participant has experienced >=Grade 2 CIT other than during the current chemotherapy treatment regimen within 6 months of Screening;
* Participant has any history of hematologic malignancies, including leukemia, myeloma, myeloproliferative disease, lymphoma, or myelodysplastic diseases;
* Participant has received >2 previous lines of chemotherapy or is receiving whole brain radiation during the study treatment period;
* Participant has a known medical history of genetic prothrombotic syndromes
* Participant has a history of arterial or venous thrombosis within 3 months of screening;
* Use of vitamin K antagonists;
* Participant has previously received a thrombopoietin receptor agonist or recombinant human thrombopoietin for the treatment of CIT within 3 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (14):
  - Dova Site, Anaheim, California
  - Dova Site, Bakersfield, California
  - Dova Site, Riverside, California
  - Dova Site, Santa Monica, California
  - Dova Site, Augusta, Georgia
  - Dova Site, Harvey, Illinois
  - Dova Site, Skokie, Illinois
  - Dova Site, Bloomington, Indiana
  - Dova Site, Wichita, Kansas
  - Dova Site, Ashland, Kentucky
  - Dova Site, Boston, Massachusetts
  - Dova Site, Minneapolis, Minnesota
  - Dova Site, Canton, Ohio
  - Dova Site, Gettysburg, Pennsylvania
- China (5):
  - Dova Site, Harbin
  - Dova Site, Linyi
  - Dova Site, Neijiang
  - Dova Site, Shanghai
  - Dova Site, Tianjin
- Hungary (4):
  - Dova Site, Budapest
  - Dova Site, Debrecen
  - Dova Site, Nyíregyháza
  - Dova Site, Törökbálint
- Poland (5):
  - Dova Site, Lublin
  - Dova Site, Olsztyn
  - Dova Site, Prabuty
  - Dova Site, Tomaszów Mazowiecki
  - Dova Site, Warsaw
- Russia (10):
  - Dova Site, Arkhangelsk
  - Dova Site, Kazan'
  - Dova Site, Kursk
  - Dova Site, Moscow
  - Dova Site, Novosibirsk
  - Dova Site, Omsk
  - Dova Site, Pyatigorsk
  - Dova Site, Saint Petersburg
  - Dova Site, Saransk
  - Dova Site, Sochi
- Serbia (3):
  - Dova Site, Belgrade
  - Dova Site, Kamenitz
  - Dova Site, Kragujevac
- Ukraine (13):
  - Dova Site, Cherkasy
  - Dova Site, Chernihiv
  - Dova Site, Chernivtsi
  - Dova Site, Ivano-Frankivsk
  - Dova Site, Kharkiv
  - Dova Site, Kherson
  - Dova Site, Kropyvnytskyi
  - Dova Site, Kyiv
  - Dova Site, Odesa
  - Dova Site, Sumy
  - Dova Site, Ternopil
  - Dova Site, Uzhhorod
  - Dova Site, Vinnytsia

REFERENCES:
- [Background] Al-Samkari H, Kolb-Sielecki J, Safina SZ, Xue X, Jamieson BD. Avatrombopag for chemotherapy-induced thrombocytopenia in patients with non-haematological malignancies: an international, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Haematol. 2022 Mar;9(3):e179-e189. doi: 10.1016/S2352-3026(22)00001-1. PMID 35240074

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 3, randomized, double- blind, placebo controlled study of the efficacy and and safety of avatrombopag in subjects with chemotherapy induced thrombocytopenia and non active non-hematologic cancers.
  The study was conducted by qualified investigators at 71 sites in China, Hungary, Poland, Russia, Serbia, Ukraine, and the United States.
  The first subject was enrolled 12October2018.
Pre-assignment Details: The study was conducted by qualified investigators at 71 sites in China, Hungary, Poland, Russia, Serbia, Ukraine, and the United States.
  The first subject was enrolled 12October2018.
Groups:
- Avatrombopag: Study is 2:1 randomization ratio (avatrombopag to placebo). 60 mg of Investigational product administered orally once daily for 5 days prior to chemotherapy and 5 days following chemotherapy treatment.
  Avatrombopag: Oral avatrombopag tablet
- Placebo: Study is 2:1 randomization ratio (avatrombopag to placebo). 60 mg Investigational product administered orally once daily for 5 days prior to chemotherapy and 5 days following chemotherapy treatment.
  Placebo Oral Tablet: Placebo comparator tablet
Period: Overall Study
Arm/Group | Avatrombopag | Placebo
Started | 82 | 40
Completed | 61 | 34
Not Completed | 21 | 6
Not completed — Withdrawal by Subject | 9 | 1
Not completed — Adverse Event | 4 | 1
Not completed — Physician Decision | 3 | 2
Not completed — Death | 2 | 0
Not completed — Other | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Avatrombopag | Placebo | Total
Number analyzed (Participants) | 82 | 40 | 122
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age at Enrollment | 61.0 (10.08) | 60.8 (10.41) | 61.0 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 22 | 65
  Male | 39 | 18 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 78 | 37 | 115
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 77 | 37 | 114
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) performance status score describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). 0=Fully active, able to carry on all pre-disease performance without restriction 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work 2=Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    Subjects with ECOG Score 0 | 21 | 8 | 29
    Subjects with ECOG Score 1 | 60 | 31 | 91
    Subjects with ECOG Score 2 | 1 | 1 | 2
Number of Eligible Chemotherapy Agents Currently Receiving per IWRS [Count of Participants; unit: Participants]
  Subjects Receiving 1 Agent | 40 | 20 | 60
  Subjects Receiving ≥ 2 Agents | 42 | 20 | 62
Baseline Platelet Count (x10⁹/L) [Mean (Standard Deviation); unit: platelets x10⁹/L] | 29.6 (13.66) | 33.0 (11.49) | 30.7 (13.04)
Height (cm) [Mean (Standard Deviation); unit: cm] | 166.3 (10.17) | 166.2 (10.32) | 166.3 (10.18)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 76.2 (17.73) | 78.8 (17.64) | 77.0 (17.67)
BMI (kg/m²) [Mean (Standard Deviation); unit: kg/m²] | 27.7 (6.56) | 28.5 (5.58) | 27.9 (6.24)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who do Not Require Platelet Transfusion, Dose Reduction in Chemotherapy by 15%, or Chemotherapy Delay by >=4 Days
Time Frame: Randomization up to 33 days
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Avatrombopag | Placebo
Number analyzed (Participants) | 82 | 40
Participants | 57 | 29
Statistical Analysis 1: Comparison: Avatrombopag vs Placebo; Test type: Other — The primary efficacy endpoint was tested between avatrombopag and placebo using the Cochran-Mantel-Haenszel 2-sided test at α=0.05, adjusting for the number of eligible chemotherapy agents as collected in IWRS (1 or ≥2 permissible chemotherapy agents); p = 0.7186, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-21.7 to 15.6]

2. Secondary Outcome: Duration of Severe Thrombocytopenia Defined as a Platelet Count <50 x 10^9/L
Description: The duration of severe thrombocytopenia is defined as the total number of days with a platelet count <50×10^9/L during the period after post-chemotherapy study drug treatment in Cycle X+1 through Chemotherapy Day of Cycle X+2.
Time Frame: Randomization up to 33 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Avatrombopag | Placebo
Number analyzed (Participants) | 81 | 40
Days | 4.6 (5.53) | 4.7 (6.56)
Statistical Analysis 1: Comparison: Avatrombopag vs Placebo; Test type: Other; p = 0.8372, Van Elteren Test

3. Secondary Outcome: Change in Platelet Count From Baseline (Nadir)
Description: Comparison of avatrombopag 60 mg vs. placebo, adjusted for the number of chemotherapy agents currently receiving per IWRS (1, ≥2).
  Cycle X nadir is defined as the lowest platelet count value prior to the first dose of study drug; Cycle X+1 nadir is defined as the lowest platelet count value during the period after post-chemotherapy study drug treatment in Cycle X+1 through Chemotherapy Day in Cycle X+2.
Time Frame: Randomization up to 33 days
Measure: Mean (Standard Deviation); unit: Platelets x 10^9/L
Arm/Group | Avatrombopag | Placebo
Number analyzed (Participants) | 82 | 40
Platelets x 10^9/L | 51.5 (61.85) | 29.1 (39.48)

4. Secondary Outcome: Percentage of Subjects Who Did Not Have Major or Non-major Clinically Relevant Bleeding During the Period After Post-chemotherapy Study Drug Treatment in Cycle X+1 Through Chemotherapy Day of Cycle X+2.
Time Frame: Randomization up to 33 days
Measure: Count of Participants; unit: Participants
Arm/Group | Avatrombopag | Placebo
Number analyzed (Participants) | 82 | 40
Participants | 82 | 40

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the Double-Blind Treatment Phase and included two 21- or 28-day chemotherapy cycles.
Description: Adverse events were assessed by Investigators at each study visit.
Arm/Group | Avatrombopag | Placebo
All-Cause Mortality (participants affected / at risk) | 2/82 | 0/40
Serious Adverse Events (participants affected / at risk) | 16/82 | 8/40
Other Adverse Events (participants affected / at risk) | 71/82 | 36/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avatrombopag (N=82) | Placebo (N=40)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 4
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Blood lactate dehydrogenase increase (Investigations) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Capillary leak syndrome (Vascular disorders) | 1 | 0
Non-small cell lung cancer (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avatrombopag (N=82) | Placebo (N=40)
Anaemia (Blood and lymphatic system disorders) | 32 | 21
Leukopenia (Blood and lymphatic system disorders) | 24 | 15
Neutropenia (Blood and lymphatic system disorders) | 24 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 15 | 13
Thombocytosis (Blood and lymphatic system disorders) | 9 | 2
Nausea (Gastrointestinal disorders) | 6 | 6
Vomiting (Gastrointestinal disorders) | 5 | 0
Asthenia (General disorders) | 5 | 4
Fatigue (General disorders) | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor will review results communications prior to public release and can embargo communications regarding trial results.

DOCUMENTS (2):
  • Study Protocol (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT03471078/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/78/NCT03471078/SAP_002.pdf